CLINICAL TRIAL: NCT03934450
Title: Metabolism and Pharmacokinetics of Primaquine Enantiomers in Human Volunteers Receiving a Seven Day Dose Regimen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Mississippi, Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PQ Study 2
Record Dates: First submitted 2018-05-14; First posted 2019-05-01 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Malaria; Glucose 6 Phosphate Dehydrogenase Deficiency
Keywords: Hemolysis; Primaquine; Pharmacokinetics
MeSH Terms: conditions — Malaria; Glucosephosphate Dehydrogenase Deficiency; Hemolysis | interventions — Primaquine

STUDY DESIGN:
Intervention Model Description: This study is a single center, prospective, cross-over phase 1 trial. Thirty-six participants will be enrolled into a two Cohort pharmacokinetic study evaluating the metabolism, pharmacokinetic behavior and tolerability of two dose levels (low/high) of primaquine enantiomers (and placebo) over the course of 7 days.
  Placebo will be added in order to assess tolerability of enantiomers. Placebo control is needed in non-drug related clinical responses.
Who Masked: Participant
Masking Description: Participants will not be able to know the sequence of the drug adminstration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RPQ (-) enantiomer (Experimental): Cohort 1 will receive 15 mg of RPQ (3A) every day for 7 days Cohort 2 will receive 22.5 mg of RPQ (3A) every day for 7 days
  Interventions: Drug: RPQ
- SPQ (+) enantiomer (Experimental): Cohort 1 will receive 15 mg of SPQ (2A) every day for 7 days Cohort 2 will receive 22.5 mg of SPQ (2A) every day for 7 days
  Interventions: Drug: SPQ
- Primaquine Phosphate (Active Comparator): Cohort 1 will receive 30 mg of RSPQ (1A) every day for 7 days Cohort 2 will receive 45 mg of RSPQ (1A) every day for 7 days
  Interventions: Drug: Primaquine Phosphate
- Placebo (Placebo Comparator): Cohort 1 will receive placebo (4A) capsules everyday for seven days Cohort 2 will receive placebo (4A) capsules everyday for seven days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RPQ — The study will compare the individual enantiomers of primaquine - R- (-)-PQ, S-(+)-PQ, and Placebo along with the racemic version.
  Other Names: R-(-) Enantiomer of Primaquine Phosphate
  Arms: RPQ (-) enantiomer
Drug: SPQ — The study will compare the individual enantiomers of primaquine - R- (-)-PQ, S-(+)-PQ, and Placebo along with the racemic version.
  Other Names: S-(+) Enantiomer of Primaquine Phosphate
  Arms: SPQ (+) enantiomer
Drug: Primaquine Phosphate — The study will compare the individual enantiomers of primaquine - R- (-)-PQ, S-(+)-PQ, and Placebo along with the racemic version.
  Other Names: Racemic Primaquine
  Arms: Primaquine Phosphate
Drug: Placebo — The study will compare the individual enantiomers of primaquine - R- (-)-PQ, S-(+)-PQ, and Placebo along with the racemic version.
  Arms: Placebo

SUMMARY:
To investigate the comparative tolerability, metabolism and pharmacokinetics of individual enantiomers of PQ in healthy human volunteers, receiving study drug over the course of 7 days.

DETAILED DESCRIPTION:
The primary objective of this project is to investigate the comparative tolerability, metabolism and pharmacokinetics of individual enantiomers of PQ in healthy human volunteers. Based on the results of this study, if one enantiomer seems to show a better safety profile (in terms of hematological effects), an analogous study will be carried out in G6PD deficient individuals (under a separate protocol). The studies are primarily aimed at understanding the tolerability and safety of the enantiomers in G6PD deficiency. If one shows a better safety profile, ultimately the evaluation of its efficacy will be required.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy adults aged 18 to 65 years

Exclusion Criteria:

* Known history of liver, kidney or hematological disease
* Known history of cardiac disease, Non Sinus Rhythm arrhythmia or QT prolongation
* Autoimmune disorders
* Report of an active infection
* Evidence of G6PD deficiency
* Participant is pregnant or breast-feeding, or is expecting to conceive during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Methemoglobin concentration in blood from baseline | Days 0, 3, 5, 7
  Change in Methemoglobin concentration in blood from baseline (% hemoglobin)

SECONDARY OUTCOMES:
Primaquine Plasma concentration, ng/mL | Days 0, 3, 5, 7
  Plasma concentrations of parent drug
Carboxy- Primaquine Plasma concentration, ng/mL | Days 0, 3, 5, 7
  Plasma concentrations of carboxy-primaquine metabolite
Primaquine N-carbamoyl-glucuronide Plasma concentration, ng/mL | Days 0, 3, 5, 7
  Plasma concentrations of Primaquine N-carbamoyl-glucuronide metabolite
Primaquine Orthoquinone Plasma concentration, ng/mL | Days 0, 3, 5, 7
  Plasma concentrations of Primaquine Orthoquinone metabolite
Change in Hematocrit (%) Compared to baseline | Days 0, 3, 5, 7
  Change in Hematocrit (%) Compared to baseline
Change in Hemoglobin (g/dL) Compared to baseline | Days 0, 3, 5, 7
  Change in Hemoglobin (g/dL) Compared to baseline
Change in AST (U/L) Compared to baseline | Days 0, 3, 5, 7
  Change in Aspartate aminotransferase (U/L) Compared to baseline; used to monitor liver function
Change in ALT (U/L) Compared to baseline | Days 0, 3, 5, 7
  Change in Alanine aminotransferase (U/L) Compared to baseline; used to monitor liver function
Change in Total Bilirubin (mg/dL) Compared to baseline | Days 0, 3, 5, 7
  Change in Total Bilirubin (mg/dL) Compared to baseline; used to monitor liver function and red cell integrity

CONTACTS AND LOCATIONS:
Overall Officials: Larry Walker, Phd, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi, University, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No